CLINICAL TRIAL: NCT00741273
Title: An Open-label, Two-stage, Dose-escalation, Parallel Group Study to Evaluate the Safety and Pharmacokinetics Profile of Proellex® (CDB-4124) in Female Patients With Impaired Hepatic Function and Healthy Adult Volunteers
Brief Title: Evaluate the Safety and PK of Proellex® in Female Patients With Impaired Hepatic Function and Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: ZP-005
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Impaired Liver Function
MeSH Terms: conditions — Liver Diseases | interventions — telapristone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proellex 25 mg healthy (Experimental): Proellex 25 mg in healthy females
  Interventions: Drug: Proellex
- Proellex 25 mg Impaired (Experimental): Proellex 50 mg in hepatically impaired females
  Interventions: Drug: Proellex

INTERVENTIONS:
Drug: Proellex — Proellex 25 mg capsule, single dose
  Other Names: Telapristone acetate

SUMMARY:
This study will evaluate the safety and pharmacokinetics of two doses of orally administered Proellex® in female patients with impaired hepatic function and healthy volunteers with normal hepatic function.

DETAILED DESCRIPTION:
16 subjects will be allocated to 2 groups. The test group will consist of 8 female patients with moderately impaired hepatic function meeting the Child-Pugh Class B severity criteria, while the control group will consist of 8 healthy female adult volunteers. During Stage I, all subjects will receive a single oral dose of 25mg of Proellex® (fasting state) and be followed in a Clinical Research Unit (CRU) for about three days. Only subjects who do not experience serious adverse events (SAEs) or adverse events (AEs) that are determined by Investigator to be possibly, probably or definitely related to the treatment will participate in Stage II. The dose will be increased to a single dose of 50mg of Proellex® (fasting state) and subjects will be followed in a Clinical Research Unit (CRU) for about three days. Subjects will undergo blood draws at several time points.

ELIGIBILITY:
Inclusion Criteria:

* Speak, read, and understand English or Spanish and is willing and able to provide written informed consent on an IRB-approved form prior to the initiation of any study procedures;
* Female, between the ages of 18 and 48 years with Body Mass Index (BMI) between 18 and 39, inclusive, are preferred; however, subjects up to 62 years old, inclusive, may participate;
* Subjects with moderate hepatic insufficiency must meet the Class B level of the Child-Pugh criteria;
* Subjects must have evidence of stable hepatic impairment;
* If on medications for treatment of the complications of liver disease, and other concomitant chronic illnesses, subjects must have been taking the medications at a stable dose for at least 10 days prior to the first dosing date and are then to be continued at the same dose for the duration of the study;
* Non-smokers are preferred, but light to moderate smoking will be allowed (no more than 10 cigarettes/day)
* Subject is willing to remain in the clinic for the screening visit and for two treatment visits (approximately 3 days for each treatment visit);
* Other inclusion criteria may apply

Exclusion Criteria:

* Past or present history of an allergic reaction to the formulations administered in this study, or in the opinion of the Investigator, suggesting an increased potential for an adverse hypersensitivity;
* Pregnant or lactating females, or women who are attempting or expecting to become pregnant at any time during the study or one month after the study;
* A physical illness within three (3) months of the study that would interfere with the study as determined by the Investigator;
* An acute illness within five (5) days of study medication administration;
* Positive urine drug screen at the screening visit based on laboratory testing;
* Other exclusion criteria may apply

Ages: 18 Years to 62 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre van As, MD, PhD, Study Director — Repros Therapeutics Inc.
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, Inc., Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy: Proellex single dose each of 25 mg and 50 mg in healthy females
- Impaired: Proellex single dose each of 25 mg and 50 mg in hepatically impaired females
Period: Overall Study
Arm/Group | Healthy | Impaired
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT and Safety populations were the same
Groups:
- Healthy: Healthy females
- Mpaired: Hepatically impaired females
- Total: Total of all reporting groups
Arm/Group | Healthy | Mpaired | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (4.1) | 54.1 (4.8) | 47.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Maximum Blood Concentration (Cmax)
Description: Cmax of a single dose of 25mg and 50mg of Proellex® in female patients with impaired hepatic function and in volunteers with normal hepatic function, assessed from samples collected at: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 5, 7, 9, 12, 16, 20, 24, 32, 36, 40 and 48 hours post dose..
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: ng/L
Groups:
- Proellex 50 mg Healthy: Proellex 50 mg in healthy females
  Proellex: Proellex 50 mg capsule, single dose
- Proellex 50 mg Impaired: Proellex 50 mg in impaired females
  Proellex: Proellex 50 mg capsule, single dose
Arm/Group | Proellex 25 mg Healthy | Proellex 25 mg Impaired | Proellex 50 mg Healthy | Proellex 50 mg Impaired
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng/L | 827.5 (312.9) | 587.6 (261.3) | 1589.5 (482.3) | 974.0 (400.2)

2. Secondary Outcome: Area Under the Curve (AUC0-t) for Proellex
Description: AUC0-t of a single dose of 25mg and 50mg of Proellex® in female patients with impaired hepatic function and in volunteers with normal hepatic function, measured from samples collected at: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 5, 7, 9, 12, 16, 20, 24, 32, 36, 40 and 48 hours post dose.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: ng x min/L
Groups:
- Proellex 25 mg Impaired: Proellex 25 mg in hepatically impaired females
  Proellex: Proellex 25 mg capsule, single dose
- 50 mg Impaired: Proellex 50 mg in impaired females
  Proellex: Proellex 50 mg capsule, single dose
Arm/Group | Proellex 25 mg Healthy | Proellex 25 mg Impaired | Proellex 50 mg Healthy | 50 mg Impaired
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng x min/L | 5147.2 (2647.3) | 3603.1 (1777.2) | 9062.4 (4616.1) | 6988.6 (3289.1)

3. Primary Outcome: Proellex Half-life (T1/2)
Description: Time for Proellex concentration to decrease by half (T1/2) of a single dose of 25mg and 50mg of Proellex® in female patients with impaired hepatic function and in volunteers with normal hepatic function,measured from samples collected at: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 5, 7, 9, 12, 16, 20, 24, 32, 36, 40 and 48 hours post dose..
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Proellex 25 mg Healthy | Proellex 25 mg Impaired | Proellex 50 mg Healthy | 50 mg Impaired
Number analyzed (Participants) | 8 | 8 | 8 | 8
Hours | 24.5 (8.4) | 37.9 (18.9) | 24.2 (10.1) | 30.9 (10.8)

ADVERSE EVENTS:
Description: Adverse events are reported together in each group for exposure to both 25mg Proellex and 50 mg Proellex
Groups:
- Proellex Healthy: Proellex 25 mg and 50 mg in healthy females
  Proellex: Proellex 25 mg and 50 mg capsule, single dose each
- Proellex Impaired: Proellex 25 mg and 50 mg in hepatically impaired females
  Proellex: Proellex 25 mg and 50 mg capsule, single dose each
Arm/Group | Proellex Healthy | Proellex Impaired
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proellex Healthy (N=8) | Proellex Impaired (N=8)
Eye pruritis (Eye disorders) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights